CLINICAL TRIAL: NCT01543373
Title: Randomized Comparison Between a DES and a BMS to Assess Neointimal Coverage by OCT Evaluation
Brief Title: Optical Coherence Tomography Comparison of Neointimal Coverage Between CRE8 DES and BMS
Acronym: DEMONSTRATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CID - Carbostent & Implantable Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C21101
Record Dates: First submitted 2012-02-20; First posted 2012-03-05 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Stable Angina; Unstable Angina; NSTEMI
Keywords: Coronary artery disease; Optical Coherence Tomography; Tissue coverage; DES
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Non-ST Elevated Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRE8 arm (Experimental)
  Interventions: Device: Amphilimus Eluting Stent
- Vision/Multilik8 arm (Active Comparator)
  Interventions: Device: Bare Metal Stent

INTERVENTIONS:
Device: Amphilimus Eluting Stent — Sirolimus formulated coronary eluting stent
  Arms: CRE8 arm
Device: Bare Metal Stent — Bare metal coronary stent
  Arms: Vision/Multilik8 arm

SUMMARY:
The purpose of the study is to demonstrate the non-inferiority of Cre8 (CID) Drug Eluting Stent, studied 3 months after implant, compared to Vision/Multilink8 Bare Metal Stent (Abbott) studied at 1 month, in terms of neointimal coverage, determined by Optical Coherence Tomography (OCT), as percentage of cross-sections with RUTTS (Ratio of Uncovered to Total Stent Struts Per Cross Section) score ≤ 0.3.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Patients with symptoms of stable or unstable angina and/or presence of a positive functional test for ischemia;
* Patient is eligible for percutaneous coronary intervention (PCI) and is an acceptable candidate for surgical revascularization (CABG);
* Left ventricular ejection fraction > 30%;
* Patients presenting with at least two vessels disease requiring a staged procedure within 3 months, according to the operator judgement;
* Target de-novo lesion;
* Target lesion located in a target vessel with a diameter ranging from 2.5 to 3.75 mm;
* Target lesion diameter stenosis > 50% and < 100% by visual estimate, with a TIMI flow of >=1;
* Discrete lesion with a length ranging from 13 to 25 mm;
* The target lesion must be appropriately covered (margin of 2.5 mm on both sides of the stent) by one study stent (Cre8 or Vision/Multilink 8), according to the randomization arm;
* Patient has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Female with childbearing potential or lactating;
* Patient presenting with acute myocardial infarction with ST elevation;
* Known allergies to antiplatelets, anticoagulants, contrast media, sirolimus or cobalt chromium;
* Cerebrovascular accident within the past 6 months;
* Acute or chronic renal dysfunction (defined as creatinine greater than 2.0 mg/dl);
* Thrombocytopenia (platelet count less than 100,000/mm³);
* Known bleeding or hypercoagulable disorder;
* Currently under immunosuppressant therapy;
* Co-morbidities that could interfere with completion of study procedures, or life expectancy less than 1 year;
* Participating in another investigational drug or device trial that has not completed the primary endpoint or would interfere with the endpoints of this study;
* Patient underwent target vessel revascularization with a DES;
* Heavily calcified vessel and/or lesion which cannot be successfully predilated or imaged by OCT
* Target lesion is located or supplied by an arterial or venous bypass graft;
* Lesion located very distally, difficult to be imaged by OCT;
* Lesion located in angulated (>70°), sharp take-off vessel;
* Target lesion involving a bifurcation with a side branch ≥2.0 mm in diameter;
* Target lesion located in the left main stem;
* Ostial lesion location;
* Target lesion has TIMI 0 flow;
* Target vessel with angiographically visible thrombus or unsuitable for proper stent delivery and deployment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Ratio of Uncovered to Total Stent Struts Per Cross Section (RUTTS) score of ≤ 0.3, determined by OCT | within 3 months from index procedure
  1 month for the BMS arm; 3 months for the DES arm

SECONDARY OUTCOMES:
Percentage of malapposed stent struts | Immediately post index procedure, 1 month (BMS arm) / 3 months (DES arm)
Percentage of malapposed and uncovered stent struts | 1 month (BMS arm) / 3 months (DES arm)
Neointimal growth and neointimal thickness | 1 month (BMS arm) / 3 months (DES arm)
Angiographic in-stent and in-segment endpoints | immediately pre and post index procedure, 1 month (BMS arm) / 3 months (DES arm)
  reference vessel diameter; minimal lumen diameter; % diameter stenosis; binary restenosis; late lumen loss
Clinical composite endpoints | At 1, 3 and 12 months
  * Cardiac death/Target vessel MI/Clinically indicated TLR
  * All death/All MI/All TVR (including TLR)
Stent Thrombosis | during index procedure, immediately after index procedure, 1 month, 3 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Prati, MD, Principal Investigator — Ospedale S. Giovanni - Addolorata
Locations (6):
- Italy (5):
  - Azienda Ospedaliero - Universitaria S.Anna, Ferrara, FE
  - Policlinico Universitario "Agostino Gemelli", Roma, RM
  - Azienda Ospedaliera S. Giovanni - Addolorata, Roma, RM
  - Presidio Ospedaliero Umberto I - Azienda Ospedaliera "Ordine Mauriziano di Torino", Torino, TO
  - ULSS n°3 - Ospedale Civile, Bassano del Grappa, VI
- University Medical Centre Utrecht, Utrecht, Netherlands